CLINICAL TRIAL: NCT00004197
Title: A Phase II Trial to Evaluate the Rate of Immune Response Using Idiotype Immunotherapies Produced by Molecular Biological Means for Treatment of Aggressive B Cell Lymphoma
Brief Title: Vaccine Therapy Plus Sargramostim Following Chemotherapy in Previously Untreated Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 0197-99-FB; P30CA036727 (NIH); GENITOPE-9902 (Other Grant/Funding Number: Genitope Corporation); SUMC-9902 (Other Grant/Funding Number: Supplemental UNMC)
Record Dates: First submitted 2000-01-21; First posted 2004-06-25 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Lymphoma
Keywords: stage I grade 3 follicular lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Mantle-Cell | interventions — keyhole-limpet hemocyanin; sargramostim; Cyclophosphamide; Doxorubicin; liposomal doxorubicin; Mitoxantrone; Prednisone; Vincristine

INTERVENTIONS:
Biological: keyhole limpet hemocyanin
Biological: sargramostim
Biological: tumor cell-based vaccine therapy
Drug: cyclophosphamide
  Other Names: Cytoxan
Drug: doxorubicin hydrochloride
  Other Names: Lipodox, Lipodox 50, and Doxil
Drug: mitoxantrone hydrochloride
  Other Names: Novantrone
Drug: prednisone
  Other Names: Prednisone Intensol, Deltasone, Rayos
Drug: vincristine sulfate
  Other Names: Kyocristine, Vincrisul, Onkovin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Vaccines may make the body build an immune response to kill cancer cells. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial of vaccine therapy plus sargramostim following chemotherapy in treating patients who have previously untreated aggressive non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the ability of recombinant idiotype immunotherapy to stimulate a specific immune response against the B cell idiotype of the malignant clone that constitutes the tumor in patients with previously untreated aggressive non-Hodgkin's lymphoma. II. Determine the safety and toxicity of this treatment regimen using Genitope Corporation's molecular rescue technology in this patient population.

OUTLINE: Patients receive induction chemotherapy consisting of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) or cyclophosphamide, mitoxantrone, vincristine, and prednisone (CNOP). Treatment repeats every 3 weeks until the maximal clinical response is achieved followed by 2 additional courses of consolidation therapy for up to a maximum of 6 courses. At 2-6 months following completion of chemotherapy, patients achieving adequate disease response receive vaccination consisting of recombinant tumor derived immunoglobulin idiotype with keyhole limpet hemocyanin conjugate subcutaneously (SQ) followed by sargramostim (GM-CSF) SQ, each at 2 separate sites on day 1. Patients receive GM-CSF alone on days 2-4. Vaccination repeats every 4 weeks for 4 doses, followed 3 months later by the fifth and final dose. Patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter until disease progression.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed aggressive non-Hodgkin's lymphoma

  * Diffuse mixed cell
  * Diffuse large cell
  * Immunoblastic Follicular large cell with more than 50% large cells
  * Mantle cell
* Non-age adjusted International Prognostic Index 2-4
* Tumor sample safely accessible by biopsy, needle aspiration, or phlebotomy
* Must have adequate circulating lymphoma cells
* Over 18 years old
* Karnofsky 80-100%
* WBC greater than 2,500/mm3
* Platelet count greater than 100,000/mm3
* Hemoglobin at least 10 g/dL
* Bilirubin less than 2.0 mg/dL SGOT/SGPT less than 2 times normal
* Creatinine less than 2.0 mg/dL
* Fertile patients must use effective contraception during and for 6 months after the study
* At least 2 months since prior nonphysiologic doses of prednisone of greater than 20 mg or equivalent
* HIV negative

Exclusion Criteria:

* No CNS metastasis
* No other illness or condition, including innate or pharmacologic immunosuppression, that would preclude study
* No other malignancy within the last 5 years except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing/negative pregnancy test
* No prior biologic therapy for lymphoma
* No prior cytotoxic chemotherapy for lymphoma
* No prior steroids for lymphoma
* No concurrent maintenance steroids or greater than 5mg of daily prednisone or equivalent
* No prior radiotherapy for lymphoma

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-06-25 (Actual); Primary Completion 2002-01-01 (Actual); Study Completion 2003-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, MD, Study Chair — University of Nebraska
Locations (2):
- United States (2):
  - Stanford University Medical Center, Stanford, California
  - University of Nebraska Medical Center, Omaha, Nebraska